CLINICAL TRIAL: NCT00044590
Title: Parkinson's Diseases Susceptibility Genes and Pesticides
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Beate Ritz, Principal Investigator, University of California, Los Angeles
Other Study IDs: 10544-CP-001
Record Dates: First submitted 2002-09-03; First posted 2002-09-05 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Pesticides; Genetic susceptibility; Polymorphisms
MeSH Terms: conditions — Parkinson Disease; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, saliva, urine, and stool samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Patients with Parkinson's Disease
- Controls: Controls, subjects without Parkinson's Disease

SUMMARY:
Parkinson's disease (PD) occurrence is higher in rural than in urban populations of industrialized countries. Epidemiologic and human tissue studies suggest that pesticides may be responsible for causing dopaminergic cell death at increased rates. While many pathophysiologic pathways may be involved in the neurodegeneration responsible for PD, genetic factors are likely to determine a general susceptibility to neurodegeneration.

DETAILED DESCRIPTION:
While many pathophysiologic pathways may be involved in the neurodegeneration responsible for PD, genetic factors are likely to determine a general susceptibility to neurodegeneration. There are a number of genetic polymorphisms of genes such as those coding for the cytochrome p450 super-family of genes referred to as 'susceptibility genes'. However, they are generally not sufficient to cause disease unless a person encounters exposure to an environmental toxin: the disease is caused by a gene-environment interaction. Thus, it is imperative to assess genetic susceptibility in individuals exposed to a toxin. We will test the gene-environment interaction hypothesis by conducting an epidemiologic population-based case-control study of newly diagnosed PD patients from three rural California counties: Kern, Fresno, and Tulare. Over a four year period, we expect to collect 400 cases referred to us by local neurologists, farm worker clinics, and Parkinson's foundations. For each case, one population control will be selected at random from residential parcel maps and Medicare databases and, in addition, one unaffected sibling control and - when possible - affected siblings to avoid potential biases and inefficiencies inherent in the use of each type of control. For each study subject, an environmental and occupational pesticide exposure estimate will be derived using California pesticide-use reporting (PUR) data and information about pesticide application on crops in combination with crop patterns shown in satellite images and aerial photographs; in addition, extensive exposure interviews will be conducted with all study subjects. In a three-tiered approach to examine the effects of gene-environment interactions we will: 1) test for association (and linkage) of PD to selected loci associated with PD in earlier studies using multiallelic repeat markers and genotyping; 2) test for association using intragenic single nucleotide polymorphisms (SNPs) of 50 candidate genes arrayed to create "the PD array"; and 3) use future technical possibilities to screen for genome wide associations using array technology to scan 5,000-10,000 SNPs throughout the genome. Data analysis will employ hierarchical modeling procedures to take into account multiple comparison issues and to incorporate prior knowledge such as increased neurotoxicity due to the interaction of gene products and chemicals.

ELIGIBILITY:
Case population inclusion criteria:

* first Parkinson's disease (PD) diagnosis after January 1998
* currently living in one of the three target counties (Kern, Tulare, Fresno)
* have lived in California for at least 5 years

Case population exclusion criteria:

* have not been diagnosed with idiopathic PD
* first PD diagnosis before January 1998
* currently living outside of Kern, Tulare, or Fresno counties
* have lived in California for fewer than 5 years

Control population inclusion criteria:

* have never been diagnosed with PD
* currently living in one of the three target counties (Kern, Tulare, Fresno)
* have lived in California for at least 5 years

Control population exclusion criteria:

* have been diagnosed with PD
* currently living outside of Kern, Tulare, or Fresno counties
* have lived in California for fewer than 5 years

For each patient, one or more unaffected sibling controls and one population control will be recruited. The population control are being selected randomly from Medicare records (95% of all controls) and residential parcel listings (for those patients younger than 65 years of age only). The controls are being marginally matched to cases according to 5-year age categories (e.g. 50-54, 55-59, 60-64, etc.), race (white, African-American, Asian, Hispanic, other), and sex. All study cases by definition will be patients who elicited care from health care providers. We are aiming to enroll every newly diagnosed PD patient into our study and expect patient population participating in our study that is as diverse as the rural population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our case population consists of patients with newly diagnosed idiopathic Parkinson's disease living in central California; they will be patients who have elicited care from health care providers. Controls will be randomly selected from Medicare records and matched to cases according to age, race, and sex.
Sampling Method: Non-Probability Sample
Enrollment: 1870 (Actual)
Dates: Start 2000-09-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beate Ritz, MD, PhD, Principal Investigator — UCLA Department of Epidemiology
Locations (1):
- Beate Ritz, UCLA Department of Epidemiology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided